CLINICAL TRIAL: NCT00043927
Title: An Open-Label, Multicenter, Randomized, Phase III Study Comparing Oral Topotecan/Cisplatin Versus Etoposide/Cisplatin as Treatment for Chemotherapy-naive Patients With Extensive Disease-Small Cell Lung Cancer.
Brief Title: Extensive Small Cell Lung Cancer Treatment Using An Investigational Drug Plus Chemotherapy In Chemotherapy-Naive Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 104864-A/389
Record Dates: First submitted 2002-08-14; First posted 2002-08-16 (Estimated); Last update posted 2013-08-21 (Estimated); Status verified 2013-08

CONDITIONS: Small Cell Lung Cancer
Keywords: Chemotherapy-naive; Small Cell Lung Cancer; SCLC; Extensive disease; ED; topotecan; Hycamtin; oral
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan; Cisplatin; PE regimen

INTERVENTIONS:
Drug: topotecan/cisplatin
Drug: etoposide/cisplatin

SUMMARY:
This study will gather and compare data about the effectiveness and safety of two different treatments for extensive Small Cell Lung Cancer (SCLC) in patients who have not received previous chemotherapy. One treatment will use an investigational drug in combination with an FDA approved chemotherapy. The other treatment will use a combination of two FDA approved chemotherapy drugs.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent (patient's written understanding of and agreement to participate in this study).
* Patients with confirmed extensive small cell lung cancer (SCLC).
* No prior chemotherapy within 5 years of the diagnosis of SCLC.
* Presence of either measurable or non-measurable SCLC by X-ray or physical examination.
* At least 3 weeks since last major surgery (a lesser period is acceptable if decided to be in the best interest of the patient).
* At least 24 hours since prior radiotherapy. Patients who have received radiotherapy must have recovered from any reversible side effects, such as nausea and vomiting.
* Laboratory criteria: Patients must have adequate bone marrow reserve and adequate kidney and liver function.

Exclusion Criteria:

* Symptoms of spreading of the disease to the brain that requires treatment with drugs called steroids.
* Any active infection.
* Severe medical problems other than the diagnosis of SCLC, that would limit the ability of the patient to follow study guidelines or that would expose the patient to extreme risk.
* Ongoing or planned chemotherapy, immunotherapy, radiotherapy, or investigational therapy for the treatment of SCLC.
* Use of an investigational drug within 30 days before the first dose of study medication.
* Women who are pregnant or lactating.
* Patients of child-bearing potential who refuse to practice an adequate form of birth control.
* Patients with clinical evidence of any stomach or intestinal (GI) condition.
* Patients requiring treatment with the drug cyclosporin A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760
Dates: Start 2001-04; Primary Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Overall Survival

SECONDARY OUTCOMES:
response rates, response duration, time to progression, tolerability and patient-perceived disease status and well being for patients

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trial, MD, Study Director — GlaxoSmithKline
Locations (157):
- United States (60):
  - GSK Clinical Trials Call Center, Hoover, Alabama
  - GSK Clinical Trials Call Center, Chula Vista, California
  - GSK Clinical Trials Call Center, Fountain Valley, California
  - GSK Clinical Trials Call Center, Greenbrae, California
  - GSK Clinical Trials Call Center, Poway, California
  - GSK Clinical Trials Call Center, Rancho Mirage, California
  - GSK Clinical Trials Call Center, Sacramento, California
  - GSK Clinical Trials Call Center, San Diego, California
  - GSK Clinical Trials Call Center, Soquel, California
  - GSK Clinical Trials Call Center, Vista, California
  - GSK Clinical Trials Call Center, Colorado Springs, Colorado
  - GSK Clinical Trials Call Center, Norwich, Connecticut
  - GSK Clinical Trials Call Center, Washington D.C., District of Columbia
  - GSK Clinical Trials Call Center, Gainesville, Florida
  - GSK Clinical Trials Call Center, Miami Shores, Florida
  - GSK Clinical Trials Call Center, Ocala, Florida
  - GSK Clinical Trials Call Center, Pensacola, Florida
  - GSK Clinical Trials Call Center, Tarpon Springs, Florida
  - GSK Clinical Trials Call Center, Atlanta, Georgia
  - GSK Clinical Trials Call Center, Augusta, Georgia
  - GSK Clinical Trials Call Center, Cumming, Georgia
  - GSK Clinical Trials Call Center, Decatur, Georgia
  - GSK Clinical Trials Call Center, Aurora, Illinois
  - GSK Clinical Trials Call Center, Chicago, Illinois
  - GSK Clinical Trials Call Center, Elk Grove Village, Illinois
  - GSK Clinical Trials Call Center, Park Ridge, Illinois
  - GSK Clinical Trials Call Center, Evansville, Indiana
  - GSK Clinical Trials Call Center, South Bend, Indiana
  - GSK Clinical Trials Call Center, New Orleans, Louisiana
  - GSK Clinical Trials Call Center, Shreveport, Louisiana
  - GSK Clinical Trials Call Center, Frederick, Maryland
  - GSK Clinical Trials Call Center, Pittsfield, Massachusetts
  - GSK Clinical Trials Call Center, Minneapolis, Minnesota
  - GSK Clinical Trials Call Center, St Louis, Missouri
  - GSK Clinical Trials Call Center, Reno, Nevada
  - GSK Clinical Trials Call Center, Voorhees Township, New Jersey
  - GSK Clinical Trials Call Center, Albuquerque, New Mexico
  - GSK Clinical Trials Call Center, Albany, New York
  - GSK Clinical Trials Call Center, New York, New York
  - GSK Clinical Trials Call Center, Rochester, New York
  - GSK Clinical Trials Call Center, Valhalla, New York
  - GSK Clinical Trials Call Center, Bismarck, North Dakota
  - GSK Clinical Trials Call Center, Cleveland, Ohio
  - GSK Clinical Trials Call Center, Columbus, Ohio
  - GSK Clinical Trials Call Center, Portland, Oregon
  - GSK Clinical Trials Call Center, Lemoyne, Pennsylvania
  - GSK Clinical Trials Call Center, Limerick, Pennsylvania
  - GSK Clinical Trials Call Center, Philadelphia, Pennsylvania
  - GSK Clinical Trials Call Center, Columbia, South Carolina
  - GSK Clinical Trials Call Center, Spartanburg, South Carolina
  - GSK Clinical Trials Call Center, Memphis, Tennessee
  - GSK Clinical Trials Call Center, Fort Worth, Texas
  - GSK Clinical Trials Call Center, Houston, Texas
  - GSK Clinical Trials Call Center, Abingdon, Virginia
  - GSK Clinical Trials Call Center, Norfolk, Virginia
  - GSK Clinical Trials Call Center, Olympia, Washington
  - GSK Clinical Trials Call Center, Yakima, Washington
  - GSK Clinical Trials Call Center, Morgantown, West Virginia
  - GSK Clinical Trials Call Center, Madison, Wisconsin
  - GSK Clinical Trials Call Center, Laramie, Wyoming
- GSK Clinical Trials Call Center, Vienna, Vienna, Austria
- Belgium (6):
  - GSK Clinical Trials Call Center, Charleroi
  - GSK Clinical Trials Call Center, Edegem
  - GSK Clinical Trials Call Center, Haine-Saint-Paul
  - GSK Clinical Trials Call Center, Leuven
  - GSK Clinical Trials Call Center, Liège
  - GSK Clinical Trials Call Center, Luxembourg
- Brazil (7):
  - GSK Clinical Trials Call Center, Belo Horizonte
  - GSK Clinical Trials Call Center, Caxias do Sul
  - GSK Clinical Trials Call Center, Fortaleza
  - GSK Clinical Trials Call Center, Porto Alegre
  - GSK Clinical Trials Call Center, Rio de Janeiro
  - GSK Clinical Trials Call Center, Salvador
  - GSK Clinical Trials Call Center, São Paulo
- Bulgaria (4):
  - GSK Clinical Trials Call Center, Burgas
  - GSK Clinical Trials Call Center, Plovdiv
  - GSK Clinical Trials Call Center, Sofia
  - GSK Clinical Trials Call Center, Varna
- Canada (15):
  - GSK Clinical Trials Call Center, Calgary, Alberta
  - GSK Clinical Trials Call Center, Edmonton, Alberta
  - GSK Clinical Trials Call Center, Winnipeg, Manitoba
  - GSK Clinical Trials Call Center, Sydney, Nova Scotia
  - GSK Clinical Trials Call Center, Newmarket, Ontario
  - GSK Clinical Trials Call Center, Oshawa, Ontario
  - GSK Clinical Trials Call Center, Ottawa, Ontario
  - GSK Clinical Trials Call Center, Peterborough, Ontario
  - GSK Clinical Trials Call Center, Sault Ste. Marie, Ontario
  - GSK Clinical Trials Call Center, Thunder Bay, Ontario
  - GSK Clinical Trials Call Center, Toronto, Ontario
  - GSK Clinical Trials Call Center, Weston, Ontario
  - GSK Clinical Trials Call Center, Greenfield Park, Quebec
  - GSK Clinical Trials Call Center, Montreal, Quebec
  - GSK Clinical Trials Call Center, Sainte-Foy, Quebec
- GSK Clinical Trials Call Center, Santiago, Chile
- China (4):
  - GSK Clinical Trials Call Center, Beijing
  - GSK Clinical Trials Call Center, Shanghai
  - GSK Clinical Trials Call Center, Wangfujing
  - GSK Clinical Trials Call Center, Xi'an
- GSK Clinical Trials Call Center, San José, Costa Rica
- Czechia (4):
  - GSK Clinical Trials Call Center, Hradec Králové
  - GSK Clinical Trials Call Center, Olomouc
  - GSK Clinical Trials Call Center, Pilsen
  - GSK Clinical Trials Call Center, Prague
- GSK Clinical Trials Call Center, Tallinn, Estonia
- Finland (3):
  - GSK Clinical Trials Call Center, Helsinki
  - GSK Clinical Trials Call Center, Kangasala
  - GSK Clinical Trials Call Center, Oulu
- France (4):
  - GSK Clinical Trials Call Center, Caen
  - GSK Clinical Trials Call Center, Calais
  - GSK Clinical Trials Call Center, Strasbourg
  - GSK Clinical Trials Call Center, Vesoul
- Germany (4):
  - GSK Clinical Trials Call Center, Heidelberg, Baden-Wurttemberg
  - GSK Clinical Trials Call Center, Ebensfeld, Bavaria
  - GSK Clinical Trials Call Center, Gauting, Bavaria
  - GSK Clinical Trials Call Center, Großhansdorf
- GSK Clinical Trials Call Center, Tegucigalpa, Honduras
- Hungary (2):
  - GSK Clinical Trials Call Center, Budapest
  - GSK Clinical Trials Call Center, Hungary
- Italy (3):
  - GSK Clinical Trials Call Center, Genoa, Liguria
  - GSK Clinical Trials Call Center, Lazio
  - GSK Clinical Trials Call Center, Roma
- GSK Clinical Trials Call Center, Kingston, Jamaica
- Lithuania (2):
  - GSK Clinical Trials Call Center, Kaunas
  - GSK Clinical Trials Call Center, Vilnius
- Mexico (3):
  - GSK Clinical Trials Call Center, Chihuahua City
  - GSK Clinical Trials Call Center, Guadalajara
  - GSK Clinical Trials Call Center, Mexico City
- Netherlands (5):
  - GSK Clinical Trials Call Center, Apeldoorn
  - GSK Clinical Trials Call Center, Arnhem
  - GSK Clinical Trials Call Center, Ede
  - GSK Clinical Trials Call Center, Harderwijk
  - GSK Clinical Trials Call Center, Nieuwegein
- New Zealand (2):
  - GSK Clinical Trials Call Center, Hamilton
  - GSK Clinical Trials Call Center, Wellington South
- GSK Clinical Trials Call Center, Oslo, Norway
- GSK Clinical Trials Call Center, Panama City, Panama
- Poland (2):
  - GSK Clinical Trials Call Center, Gdansk
  - GSK Clinical Trials Call Center, Kielce
- GSK Clinical Trials Call Center, Ponce, Puerto Rico
- Russia (2):
  - GSK Clinical Trials Call Center, Moscow
  - GSK Clinical Trials Call Center, Moscow Region
- GSK Clinical Trials Call Center, Singapore, Singapore
- Slovakia (4):
  - GSK Clinical Trials Call Center, Banská Bystrica
  - GSK Clinical Trials Call Center, Bratislava
  - GSK Clinical Trials Call Center, Košice
  - GSK Clinical Trials Call Center, Nitra
- GSK Clinical Trials Call Center, Johannesburg, Gauteng, South Africa
- GSK Clinical Trials Call Center, Seoul, South Korea
- Spain (2):
  - GSK Clinical Trials Call Center, Valencia, Valencia
  - GSK Clinical Trials Call Center, Lleida
- GSK Clinical Trials Call Center, Taipei, Taiwan
- United Kingdom (6):
  - GSK Clinical Trials Call Center, Aberdeen, Aberdeenshire
  - GSK Clinical Trials Call Center, Nottingham, Nottinghamshire
  - GSK Clinical Trials Call Center, Glasgow
  - GSK Clinical Trials Call Center, Leeds
  - GSK Clinical Trials Call Center, Leicester
  - GSK Clinical Trials Call Center, Poole